CLINICAL TRIAL: NCT02962674
Title: ProstaCare Water Electrolysis System for the Treatment of Benign Prostatic Hyperplasia
Brief Title: To Evaluate the Safety and Performance of the ProstaCare Water Electrolysis System in Relieving Symptoms of BPH.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: ProstaCare Singapore Pte. Ltd. (Industry)
Responsible Party: Sponsor
Organization: ProstaCare Pty Ltd (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP# PC 1.0
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Results first posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: BPH
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Other)
  Interventions: Device: prostaFix System

INTERVENTIONS:
Device: prostaFix System

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the ProstaCare System in relieving symptoms of urinary outflow obstruction secondary to benign prostatic hyperplasia.

ELIGIBILITY:
Key Inclusion Criteria:

* 45 years of age or older with a diagnosis of BPH,
* International Prostate Symptom Score (IPSS) of 12 or greater,
* Prostate volume between 25 cm3 and 55 cm3,
* Uroflow with peak flow rate (Qmax) no greater than 13 ml/sec with a corresponding voided volume of at least 100 ml and a post void residual (PVR) of 250 ml or less.
* Prostate length, width and height must be at least 3.2 cm, 3.5 cm and 2.5 cm, respectively

Key Exclusion Criteria:

* Obstruction due to an enlarged middle lobe, central gland or significant transverse asymmetry,
* Subjects on 5 alpha reductase inhibitors (5-ARI) (inclusion only if washed out prior to treatment),
* Subjects on alpha blockers (inclusion only if washed-out before treatment),
* Active urinary tract infection at time of treatment,
* Interest in maintaining fertility,
* Past history of urologic surgery or minimally invasive treatment for BPH,
* History of or current medical conditions contraindicating elective urological procedures.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2020-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Ho Sun Sien, MD, Principal Investigator — Singapore General Hospital
Locations (3):
- Urology Bay of Plenty (BOP), Tauranga, New Zealand
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- prostaFix System: Subjects treated with the prostaFix Water Electrolysis System
Period: Overall Study
Arm/Group | prostaFix System
Started (All subjects that signed an informed consent form.) | 49 (Although a total of 49 subjects were consented to participate in the study, three (3) of those subjects are not included in the study analysis as they did not actually receive treatment. These 3 subjects could not be treated because of their anatomy and therefore are considered "treatment attempts". The final enrollment number (treated subjects only)is 46 subjects.)
3 Month Endpoint | 46 (All treated subjects that completed the 3-month endpoint visit per protocol.)
12 Month Durability | 46 (All subjects that completed the 12-month follow-up visit per protocol.)
24 Month Durability | 32 (All subjects that completed the 24-month follow-up visit. Note that at the time of study termination, all subjects would have reached this milestone.)
36 Month Durability | 18 (All subjects that completed the 36-month follow-up visit. Note that at the time of study termination, not all subjects would have reached this milestone depending on time of enrollment.)
48 Month Durability | 4 (All subjects that completed the 48-month follow-up visit. Note that at the time of study termination, not all subjects would have reached this milestone depending on time of enrollment.)
Completed | 0 (Study was terminated by sponsor prior to reaching 60 Month study completion mainly due to COVID-19 effects on subject follow-up.)
Not Completed | 49
Not completed — Study terminated by sponsor prior to completion of all study protocol visits by enrolled subjects. | 49

BASELINE CHARACTERISTICS:
Population: All subjects who enrolled in the study and were treated with the prostaFix System.
Groups:
- Treatment: Subjects treated with the prostaFix System
Arm/Group | Treatment
Number analyzed (Participants) | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Chinese | 28
  Race: Malay | 2
  Race: Indian | 2
  Race: New Zealand European | 14
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 14
  Singapore | 32

OUTCOME MEASURES:

1. Primary Outcome: Mean International Prostate Symptom Score (IPSS) at 3 Months Follow-up Visit
Description: The primary effectiveness objective was to demonstrate that mean IPSS improvement (Δ IPSS) following treatment with the prostaFix System exceeded 6.5 points with 95% confidence 3 months after treatment.
  The International Prostate Symptom Score (IPSS) is a validated questionnaire used to assess baseline and post treatment BPH symptoms. It is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the subject to choose one out of six answers indicating increasing severity of that particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic): Mild (symptom score less than or equal to 7), Moderate (symptom score range 8-19) and Severe (symptom score range 20-35). Improvement in BPH symptoms is seen as a decrease in IPSS.
Time Frame: 3 months after treatment
Population: Intent-to-treat (ITT) with last observation carried forward (LOCF): All subjects who enrolled in the study, were treated with the prostaFix System, and completed the 3 month follow-up visit without significant protocol deviations.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | prostaFix System
Number analyzed (Participants) | 46
score on a scale | 12.3 (1.22)
Statistical Analysis 1: Comparison: prostaFix System; The null and alternative hypotheses associated with this objective was written as: H0: μ ΔIPSS ≤ 6.5 points HA: μ ΔIPSS > 6.5 points where μ ΔIPSS was the true underlying value of mean ΔIPSS following a treatment at the 3-month follow-up visit and 6.5 points was an objective performance goal (OPG). The objective was met at a given time point by rejecting the null hypothesis in a one-sided t-test at the 5% significance level; Test type: Superiority; p = 0.004, t-test, 1 sided

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: The primary safety objective of this study was to estimate the proportion of subjects affected by serious adverse events (SAEs) associated with the use of the device. This objective was addressed through recording all adverse events (AEs) observed or reported during the course of the study.
Time Frame: 3 months after treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | prostaFix System
Number analyzed (Participants) | 46
Participants | 0

3. Secondary Outcome: Mean Change in QOL From Baseline
Description: Question eight of the IPSS questionnaire refers to the subject's perceived quality of life (QOL). The International Scientific Committee (SCI), under the patronage of the World Health Organization (WHO) and the International Union Against Cancer (UICC), recommends the use of only a single question to assess the quality of life. The answers to this question range from "delighted" to "terrible" or 0 to 6.
Time Frame: Baseline and 3 months after treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | prostaFix System
Number analyzed (Participants) | 46
score on a scale | -2.2 (0.25)

4. Secondary Outcome: Mean Change in Peak Flow Rate (Qmax) From Baseline
Description: Uroflowmetry measures the flow of urine. It tracks how fast urine flows (peak flow rate - Qmax), how much flows out, and how long it takes. It's a diagnostic test to assess how well the urinary tract functions. Uroflowmetry is used in BPH subjects to help the doctors determine how well the subject's urinary tract is doing and the severity of obstruction caused by the prostate. The higher the Qmax is, the less obstructed the urethra.
Time Frame: Baseline and 3 months after treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ml/sec
Arm/Group | prostaFix System
Number analyzed (Participants) | 46
ml/sec | 2.36 (0.64)

5. Secondary Outcome: Mean Change in Post Void Residual (PVR) From Baseline
Description: The Post Void Residual (PVR) is an indicator of urine remaining in the bladder after voiding. A healthy bladder should be fairly empty following urination. A volume < 50 mL is normal; < 100 mL is usually acceptable in patients > 65 years old. The higher the PVR, the more urine is left in the bladder and this can be seen as a sign of increased obstruction of the urethra.
Time Frame: Baseline and 3 months after treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ml
Arm/Group | prostaFix System
Number analyzed (Participants) | 46
ml | -3.54 (9.46)

6. Secondary Outcome: Mean Change in MSHQ-EjD Score From Baseline
Description: The MSHQ-EjD Short Form (Male Sexual Health Questionnaire - Ejaculatory Disfunction) is composed of three questions that rate ejaculatory function in men. A fourth question measures the MSHQ-EjD Bother, this asks the subject if he is bothered by his level of ejaculatory function.
  MSHQ-EjD total score ranges from 1 to 15 with a higher score indicating better sexual functioning. MSHQ-EjD bother score ranges from 0 to 5 with a higher score indicating greater bother. An increase in the MSHQ-EjD Total Score indicates better ejaculation and a decrease in the MSHQ-EjD Bother Score means that the subject is less bothered by his ejaculatory function. Due to the sensitive nature of the questions, this questionnaire is voluntary and not all subjects completed it at baseline. Some subjects completed at baseline but decided not to complete at certain follow-up visits which explains the different number of participants during various analysis time frames.
Time Frame: Baseline and 3 months after treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | prostaFix System
Number analyzed (Participants) | 46
score on a scale
  MSHQ-EjD (Total): number analyzed (Participants) | 28
  MSHQ-EjD (Total) | 0.6 (0.48)
  MSHQ-EjD (Bother): number analyzed (Participants) | 29
  MSHQ-EjD (Bother) | -0.4 (0.32)

7. Secondary Outcome: Change in IIEF Score From Baseline
Description: The IIEF (International Index of Erectile Function) provides a broad measure of sexual function; an increase in score indicates an improvement in sexual function. This questionnaire consists of five questions that asks the subject of any erection problems that have impacted his sexual life over the past 4 weeks or since the last study visit, whichever is shorter. IIEF total score ranges from 0 to 25 with a higher score indicating better sexual functioning and an increase in score indicates an improvement in sexual function. Due to the sensitive nature of the questions, this questionnaire is voluntary and not all subjects completed it at baseline. Some subjects completed at baseline but decided not to complete at certain follow-up visits which explains the different number of participants during various analysis time frames.
Time Frame: Baseline and 3 months after treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | prostaFix System
Number analyzed (Participants) | 30
score on a scale | -0.5 (1.12)

8. Secondary Outcome: Mean Change in IPSS From Baseline
Description: The International Prostate Symptom Score (IPSS) is a validated questionnaire used to assess baseline and post treatment BPH symptoms. It is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the subject to choose one out of six answers indicating increasing severity of that particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic): Mild (symptom score less than or equal to 7), Moderate (symptom score range 8-19) and Severe (symptom score range 20-35). Improvement in BPH symptoms is seen as a decrease in IPSS.
Time Frame: Baseline and 12 months from treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | prostaFix System
Number analyzed (Participants) | 46
score on a scale | -8.6 (1.06)

9. Secondary Outcome: Mean Change in QOL From Baseline
Description: as for outcome 3
Time Frame: Baseline and 12 months from treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | prostaFix System
Number analyzed (Participants) | 46
score on a scale | -1.3 (0.20)

10. Secondary Outcome: Mean Change in Peak Flow Rate (Qmax) From Baseline
Description: as for outcome 4
Time Frame: Baseline and 12 months from treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ml/sec
Arm/Group | prostaFix System
Number analyzed (Participants) | 46
ml/sec | 0.99 (0.49)

11. Secondary Outcome: Mean Change in Post Void Residual (PVR) From Baseline
Description: as for outcome 5
Time Frame: Baseline and 12 months from treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ml
Groups:
- protaFix System: Subjects treated with the prostaFix Water Electrolysis System
Arm/Group | protaFix System
Number analyzed (Participants) | 46
ml | -1.82 (9.64)

12. Secondary Outcome: Mean Change in MSHQ-EjD From Baseline
Description: as for outcome 6
Time Frame: Baseline and 12 months from treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | prostaFix System
Number analyzed (Participants) | 46
score on a scale
  MSHQ-EjD (Total): number analyzed (Participants) | 28
  MSHQ-EjD (Total) | -0.6 (0.5)
  MSHQ-EjD (Bother): number analyzed (Participants) | 29
  MSHQ-EjD (Bother) | -0.2 (0.34)

13. Secondary Outcome: Mean Change in IIEF From Baseline
Description: as for outcome 7
Time Frame: Baseline and 12 months from treatment
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 30
score on a scale | -1.9 (1.23)

14. Secondary Outcome: MRI Necrosis Volume
Description: The prostaFix System uses pH shifts induced by water electrolysis to induce necrosis in the hyperplastic prostate tissue. The induced necrosis within the borders of the prostate result in a pressure reduction and thereby relieve the symptoms of BPH. This necrosis that resulted from the procedure eventually heals and necrosis volume should reduce overtime. Per protocol, only the first 10-15 subjects would have MRI studies at done to assess subject safety and treatment effect. then MRI was optional. A total of 14 subjects actually had an MRI and the results are reported for those subjects.
Time Frame: 3 months after treatment
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | prostaFix System
Number analyzed (Participants) | 14
cm^3 | 0.12 (0.25)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment until study termination. All enrolled subjects were followed to at least their 12-month follow-up visit.
Description: AEs were classified by the investigator at each corresponding site for relatedness to the device and seriousness based on the Common Terminology Criteria for Adverse Events (Version 4.03) (CTCAE) (US Department of Health and Human Services 2010) guidelines. In addition, the adverse events were coded using MedDRA and reviewed by the Medical Advisor.
Arm/Group | prostaFix System
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 3/46
Other Adverse Events (participants affected / at risk) | 24/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | prostaFix System (N=46)
Haematuria (Renal and urinary disorders) | 1 (1)
Haemorrhage (secondary) (Surgical and medical procedures) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | prostaFix System (N=46)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Hypertonic bladder (Renal and urinary disorders) | 6 (6)
Lower urinary tract symptoms (worsened) (Renal and urinary disorders) | 13 (13)
Urinary retention (Renal and urinary disorders) | 3 (3)
Urinary urgency (Renal and urinary disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT02962674/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/74/NCT02962674/SAP_001.pdf